CLINICAL TRIAL: NCT01398527
Title: An Interdisciplinary Knowledge Translation Intervention in Long-term Care: The Vitamin D and Osteoporosis Study (ViDOS) Pilot Cluster Randomized Controlled Trial
Brief Title: Vitamin D Osteoporosis Long-Term Care Study
Acronym: ViDOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Dr. Alexandra Papaioannou, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB 09-215
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2013-05

CONDITIONS: Osteoporosis
Keywords: Long-Term Care; Vitamin D
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LTC Osteoporosis Toolkit Only (No Intervention): Homes will receive the LTC osteoporosis toolkit only and will be required to attend an online webinar to outline the toolkit contents.
- Educ sessions & LTC Osteoporosis toolkit (Active Comparator): LTC homes will receive the LTC osteoporosis toolkit, on line webinar. Three educational sessions lead by an osteoporosis expert will also take place, 1 on-site visit and 2 webinars.

INTERVENTIONS:
Other: Educ sessions & LTC Osteoporosis toolkit — Three points of contact to be made. The first being a 1-hour personal visit at each intervention LTC home from an osteoporosis expert with the homes professional or health advisory committee (PAC or HAC). The second and third contact points will be made through webinars between the osteoporosis expert and the group from the first meeting.
  Other Names: Knowledge translation

SUMMARY:
The research question is, does a multifaceted, multidisciplinary intervention including small groups, chart audits and point of care tools, increase the number of people receiving optimal vitamin D therapy in the long term care (LTC) setting? Secondary outcomes include the number of falls and fractures experienced by the residents in each LTC home and the number of residents receiving appropriate bisphosphonate therapy.

DETAILED DESCRIPTION:
This is a cluster randomized controlled trial. In the long-term care (LTC) setting, more research is needed on how health care professionals can be kept up to date on the latest medical evidence for providing care to elderly residents. The LTC environment differs from other health care settings. We need to examine what types of strategies can be used to effectively educate LTC physicians, nurses, and other care professionals about the best care practices.

In this study, we will deliver and evaluate a multi-component educational strategy that builds on research in LTC by our team. In order to evaluate its success, 20 homes will receive the intervention and 20 homes will receive usual care. In the intervention homes, a team of experts will give educational sessions at the LTC home, delivering key messages about "best practices", helping LTC professionals to plan changes for delivering better care, giving feedback about performance, and providing materials (e.g., DVD, treatment plans). We will also train a professional in the home to "champion" the cause after the experts are gone.

The specific "best practices" topic we have chosen to test our model is osteoporosis and fractures. These conditions are very common in the elderly living in LTC and negatively impact quality of life. For example, an individual with a hip or other fracture may experience unnecessary pain and suffering and even pre-mature death. There are effective treatments that can be used to reduce fractures, including vitamin D, which is a low-cost, well-tolerated and easy treatment to deliver. Unfortunately our previous studies have shown that most LTC residents are not receiving effective fracture-prevention treatments. To determine our intervention's success, we will examine whether the rate of vitamin D use and other treatments increases, and whether fewer LTC residents fall and fracture. We are also interested in studying the strategy's format and feasibility and what future changes should be made.

ELIGIBILITY:
Inclusion Criteria:

* LTC homes in Ontario that are serviced by MPGI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of LTC residents on vitamin D | 16 months

SECONDARY OUTCOMES:
Number of falls and fractures | 16 months
Vitamin D dose | 16 months
Bisphosphonate use by LTC residents | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University - St. Peter's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Borhan S, Kennedy C, Ioannidis G, Papaioannou A, Adachi J, Thabane L. An empirical comparison of methods for analyzing over-dispersed zero-inflated count data from stratified cluster randomized trials. Contemp Clin Trials Commun. 2020 Feb 1;17:100539. doi: 10.1016/j.conctc.2020.100539. eCollection 2020 Mar. PMID 32072073
- [Derived] Kennedy CC, Ioannidis G, Thabane L, Adachi JD, Marr S, Giangregorio LM, Morin SN, Crilly RG, Josse RG, Lohfeld L, Pickard LE, van der Horst ML, Campbell G, Stroud J, Dolovich L, Sawka AM, Jain R, Nash L, Papaioannou A. Successful knowledge translation intervention in long-term care: final results from the vitamin D and osteoporosis study (ViDOS) pilot cluster randomized controlled trial. Trials. 2015 May 12;16:214. doi: 10.1186/s13063-015-0720-3. PMID 25962885
- [Derived] Kennedy CC, Thabane L, Ioannidis G, Adachi JD, Papaioannou A; ViDOS Investigators. Implementing a knowledge translation intervention in long-term care: feasibility results from the Vitamin D and Osteoporosis Study (ViDOS). J Am Med Dir Assoc. 2014 Dec;15(12):943-5. doi: 10.1016/j.jamda.2014.05.007. Epub 2014 Jun 18. PMID 24953541
- [Derived] Kennedy CC, Ioannidis G, Giangregorio LM, Adachi JD, Thabane L, Morin SN, Crilly RG, Marr S, Josse RG, Lohfeld L, Pickard LE, King S, van der Horst ML, Campbell G, Stroud J, Dolovich L, Sawka AM, Jain R, Nash L, Papaioannou A. An interdisciplinary knowledge translation intervention in long-term care: study protocol for the vitamin D and osteoporosis study (ViDOS) pilot cluster randomized controlled trial. Implement Sci. 2012 May 24;7:48. doi: 10.1186/1748-5908-7-48. PMID 22624776